CLINICAL TRIAL: NCT03437460
Title: The Economic and Cognitive Effects of Pain Reduction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Implementation issues
Sponsor: University of Pennsylvania (Other)
Collaborators: Institute for Financial Management and Research (Other)
Responsible Party: Principal Investigator, Heather Schofield, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 825454
Record Dates: First submitted 2017-07-12; First posted 2018-02-19 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Pain, Chronic
Keywords: Productivity; Cognitive Function; Decision Making; Well-Being; Health; Labor
MeSH Terms: conditions — Chronic Pain | interventions — Ibuprofen; Prenatal Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen 600mg (Active Comparator): Treatment group participants receive a single 600 mg of over-the-counter ibuprofen.
  Interventions: Drug: Ibuprofen 600 mg
- Prenatal vitamins (Placebo Comparator): The placebo group participants receive a single dose of a pre-natal multivitamin.
  Interventions: Dietary Supplement: Prenatal vitamins
- Control group (No Intervention): Control-group participants are not provided with any treatment and they are fully informed regarding their treatment status.

INTERVENTIONS:
Drug: Ibuprofen 600 mg — The investigators administer one single 600 mg dose of ibuprofen immediately before lunch. Participants are then asked to complete the cold pressor task, flower stringing sessions, and cognitive tasks.
  Other Names: Brufen
  Arms: Ibuprofen 600mg
Dietary Supplement: Prenatal vitamins — The investigators administer one single prenatal multivitamin immediately before lunch. Participants are then asked to complete the cold pressor task, flower stringing sessions, and cognitive tasks.
  Arms: Prenatal vitamins

SUMMARY:
Physical pain is a common but largely overlooked aspect of the lives of the poor. Not only does pain directly reduce life quality and happiness, it may also hamper cognitive function and, consequently, decision-making, productivity, and earnings. Workers with chronic pain may work fewer days, take longer breaks, and make less-considered choices regarding inputs; all outcomes that would reduce output and lead to greater impoverishment or impede the productivity and profitability of microenterprises and firms. The investigators will take the first steps in understanding the broader causal impact of physical pain on the cognitive and economic lives of the poor via a randomized controlled trial (RCT). 450 low-income women in Chennai, India, will be assigned to one of three treatment arms: 600 mg of over-the-counter pain medication, a placebo pill, or no medication. The research will quantify the causal impact of reduced pain on previously unstudied outcomes essential to escaping poverty including cognitive function, productivity, and earnings.

DETAILED DESCRIPTION:
The investigators propose to evaluate the effect of reductions in chronic physical pain on cognitive function and productivity among poor individuals via a simple intervention using over-the-counter (OTC) pain medication. To do this, the investigators will enroll 450 low-wage female workers in Chennai, India into a two-day randomized controlled trial in which 150 randomly selected participants will receive OTC Non-steroidal Anti-inflammatory Drugs (NSAIDs; namely, Ibuprofen) at FDA-approved levels of one dose of 600 mg each on a single day, 150 participants will receive a placebo pill, and 150 participants will serve as a no-treatment control group.

Participants will complete a detailed survey, a battery of cognitive tests, pain measurements, a task to objectively scale each participant's pain assessments, and a task designed to measure economic productivity as detailed below.

Study location:

The study will be based at the Behavioral and Development Economics Lab in Chennai, India, founded by PIs Schofield and Schilbach in conjunction with a local institution, the Institute for Financial Management and Research (IFMR).

Sample:

Participants will consist of female flower stringers in Chennai, India. Flower stringers are self-employed individuals typically working on the streets. These women purchase flowers in the morning, string them together, and sell the strands to customers passing by. Their average daily income is Rs. 250-500 (approximately $4-9). Preliminary survey evidence suggests a higher prevalence of physical pain among older individuals; hence, this study will limit enrollment to individuals aged 25 to 65 years. The investigators focus on this population for several additional reasons. First, the nature of their work (stringing flowers while sitting on the floor for most of the day) causes high levels of pain. Second, due to the societal norms in the area, women do not regularly consume significant amounts of alcohol, substantially lowering the risks associated with taking pain medication. Third, the nature of their work makes flower stringers' productivity easily measurable (length and weight of flowers strung). Finally, although this population is specific, participants are similar in many ways (e.g. age, education, labor habits) to many workers in the informal sector, improving the study's external validity.

Recruitment and screening:

Surveyors approach potential participants at their place of work (typically a stand on the side of the street). The surveyor shares information about the study, while also conducting a broad first screen for eligibility. If participants are interested in participating and pass the initial screening, they schedule a time to come in to the lab for Day 1 (see below for further detail on the timing of the study). On Day 1, all potential participants are further screened to ensure: 1) their primary profession is flower-stringing, 2) they do not have any health conditions which are contraindicated for taking ibuprofen, 3) they regularly experience pain from their work, and 4) they are between the ages of 25 and 65.

Timing:

Day 1: Following field recruitment, potential participants are screened for eligibility and complete an informed consent process. If eligible, participants complete the survey measuring demographics, work habits, and data on the type and amount of pain typically experienced. Participants also complete the battery of cognitive assessments.

The investigators will randomize using Stata and then reveal the experimental condition assignment to individuals privately. Any non-compliance will be carefully tracked.

Day 2: Participants complete the battery of cognitive tasks and 30 minutes of flower stringing in the morning (pre-treatment). Participants report their pain levels periodically and complete a "pain calibration" by reporting their pain levels while holding their hand in cold water. They are then randomly assigned to one of the three experimental arms at lunch. After lunch, all participants complete another 3 hours of flower-stringing and repeat the battery of cognitive tasks. Participants also complete a "pain tolerance test" after lunch. In this task, participants are paid for the time they leave their hand in cold water.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 25 and 65
* Must speak Tamil as their primary language
* Must report that they have suffered from chronic physical pain in the last week.

Exclusion Criteria:

* An adverse relation related to pain medication in the past
* Kidney disease (ongoing or kidney stone within the past 3 years)
* Gastrointestinal (GI) discomfort
* History of complicated peptic ulcer disease
* Currently using NSAIDs, aspirin, corticosteroids or anticoagulants
* Allergies to any of the medicines use in the study
* History of gastric bleeding
* History or existing liver disease
* Surgery within 1 to 2 weeks after the study
* Hypertension
* Heart disease or failure
* Diabetes
* Lupus
* Blood clotting
* Actual or potential pregnancy
* Use of contraindicated medications (including anticoagulants)
* Suicidal thoughts
* Consumption of more than 14 alcoholic beverages a week.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Change in pain levels - visual analog scale | Change from baseline to end of Day 2
  Visual analog scale pain levels will measure the participant's self-assessed pain levels throughout the day. On the morning of Day 2 of the study, visual analog scale pain levels are recorded after each of the 4 cognitive tasks and after 30 minutes of flower stringing. Visual analog scale pain levels are reported throughout the afternoon of study Day 2 after each cognitive task and after every 30 minutes of flower stringing, and then compared to the baseline measures.
Change in pain levels - cold pressor task | Change from baseline to end of Day 2
  Cold pressor task will measure the participant's pain tolerance. To assess a baseline tolerance, participants are asked to place their hand in cold water for 5 seconds to become accustomed to the task, and then for 20 seconds, after which they report their pain level. After lunch, participants complete the cold pressor duration, during which they hold their hand in cold water for as long as they want, up to 2 minutes. This measure is compared to the baseline measure from the morning.
Change in cognitive function: impulse control | Change from baseline to end of Day 2
  The Hearts and Flowers task is completed once in the morning as a baseline measure and twice in the afternoon, to compare to the baseline. The task is compensated according to performance.
Change in cognitive function: simple memory | Change from baseline to end of Day 2
  The Corsi block-span task is completed once in the morning as a baseline measure and twice in the afternoon, to compare to the baseline. The task is compensated according to performance.
Change in cognitive function: working memory | Change from baseline to end of Day 2
  The N-back task is completed once in the morning as a baseline measure and twice in the afternoon, to compare to the baseline. The task is compensated according to performance.
Change in cognitive function: simple attention | Change from baseline to end of Day 2
  The Psychomotor Vigilance is completed once in the morning as a baseline measure and twice in the afternoon, to compare to the baseline. The task is compensated according to performance.
Change in flower-stringing productivity: weight of flower buds used | Change from baseline to end of Day 2
  Flower stringing productivity (weight of buds used) baseline is measured in the morning after a 30 minute flower stringing session. This outcome is compared to the weight of flower buds used in the afternoon flower stringing sessions, which span 150 minutes and 30 minutes.
Change in flower-stringing productivity: length of garland | Change from baseline to end of Day 2
  Flower stringing productivity (length of garland) baseline is measured in the morning after a 30 minute flower stringing session. This outcome is compared to the length of garland in the afternoon flower stringing sessions, which span 150 minutes and 30 minutes.
Change in flower-stringing productivity: density of garland | Change from baseline to end of Day 2
  Flower stringing productivity (density of garland) baseline is measured in the morning after a 30 minute flower stringing session. This outcome is compared to the density of garland in the afternoon flower stringing sessions, which span for 150 minutes and then for 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Schilbach, Ph.D., Principal Investigator — MIT Department of Economics; Heather Schofield, Ph.D., Principal Investigator — University of Pennsylvania, Perelman School of Medicine and Wharton Business School; Anuj Shah, Ph.D., Principal Investigator — University of Chicago, Booth School of Business; Sendhil Mullainathan, Ph.D., Principal Investigator — Harvard University; Emma Dean, M.S., Principal Investigator — University of Pennsylvania, Wharton School of Business
Locations (1):
- Institute for Financial Management and Research, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to other researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available upon completion of the study with additional time to allow for merging, cleaning, and publication.
Access Criteria: Data are available upon request following publication.

DOCUMENTS (1):
  • Informed Consent Form (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03437460/ICF_000.pdf